CLINICAL TRIAL: NCT04723186
Title: Open-Label, Sequential-Dose Escalation/De-escalation Trial Testing MT1002 in Patients Undergoing PCI Due to Acute Coronary Syndrome With NSTEMI
Brief Title: MT1002 Phase II Study in ACS Patients With PCI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was decided to be terminated due to commercial considerations,（not the safety issues of the product）.
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT1002-II-C01
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-05

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS, PCI
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Open-Label, Sequential-Dose Escalation/De-escalation Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Monotherapy of MT1002, 3 doses via intravenous (IV) + infusion (Experimental): Three doses of MT1002 (IV loading + continuous IV infusion) will be sequentially tested. The first dose level is 0.90 mg/kg initial loading dose (bolus intravenous injection) + 1.8 mg/kg/h (infusion) for 4 hours. The second dose level will be based on the results from the first cohort (If the dose is escalated, then the second dose level is 1.2 mg/kg initial loading dose (bolus intravenous injection) + 2.3 mg/kg/h (infusion) for 4 hours; if the dose is de-escalated, then the second dose level is 0.6 mg/kg initial loading dose (bolus intravenous injection) + 1.2 mg/kg/h (infusion) for 4 hours). The third dose will be determined based on the results from the first 2 cohorts.
  Interventions: Drug: MT1002 for Injection

INTERVENTIONS:
Drug: MT1002 for Injection — MT1002 will be initiated as close to the start of PCI as possible. MT1002 should be initiated during diagnostics angiography when indication for PCI is confirmed, provided the PCI is indicated right after the coronary angiography. PCI can start after MT1002 initiation as soon as ACT is confirmed to be ≥ 200 sec or within 30 min after MT1002 starts, whichever occurs first. MT1002 will be administered by an intravenous injection of 0.90 mg/kg, 1.2 mg/kg, or 0.6 mg/kg (depending on the dose selected for the cohort) prior to the PCI procedure, immediately followed by an IV infusion of 1.8 mg/kg/hour, 2.3 mg/kg/hour, or 1.2 mg/kg/hour (depending on the dose selected for the cohort) until completion of the procedure. At completion of PCI, subjects will be continued on IV MT1002 for 4 hours from infusion start.

SUMMARY:
This is an open-label, sequential-dose escalation/de-escalation trial testing 3 dose levels of MT1002 in patients undergoing PCI due to ACS with NSTEMI. Three doses of MT1002 will be sequentially tested in cohorts of 6 patients each to achieve target ACT.

DETAILED DESCRIPTION:
MT1002 is a novel 32-amino acid synthetic peptide aimed to combine molecular functions of both a direct thrombin inhibitor and a platelet glycoprotein IIb/IIIa receptor antagonist, indicated for use as an antithrombotic and anticoagulant in patients with ACS and in patients undergoing PCI. This study is to investigate the safety, tolerability, and efficacy of MT1002 in patients undergoing PCI due to ACS with NSTEMI.

This study is a single dose, sequential-dose escalation study in patients undergoing PCI due to ACS with NSTEMI. The first 2 doses were considered safe and well tolerated in the Phase 1 healthy subject study. The third dose to be given will be determined based on the safety and efficacy results from the first 2 doses. Dose escalation/de-escalation and stopping rules have been put in place to ensure the safety of the patients in this study.

The patients will receive a single MT1002 close to the initiation of PCI (Day 1) followed by 4 hours of IV infusion and follow-up at Day 2, Day 14, and Day 30.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 to 85 years of age.
2. Diagnosed with NSTEMI.
3. Patients who will undergo PCI during the index hospitalization for an NSTEMI.
4. Ability to understand and willing to give written informed consent.
5. Women of childbearing potential must have a negative pregnancy test or be post-menopausal for at least 1 year before enrollment or be permanently sterilized since ≥6 weeks. Females of childbearing potential and males with partners of childbearing potential must be using effective contraception.

Exclusion Criteria:

1. .Cardiogenic shock or prolonged cardiopulmonary resuscitation (CPR).
2. Active bleeding, bleeding diathesis, coagulopathy.
3. Any history of intracranial bleeding or structural abnormalities.
4. Prior transient ischemic attack, prior stroke within 6 months.
5. Index MI is STEMI or new left bundle branch block.
6. The following planned procedures within 30 days after enrollment: staged PCI, CABG, valve surgery, or additional invasive procedures.
7. Pre-existing atrial fibrillation or prolonged QTcF (470ms in men, 480ms in women).
8. Anticipated requirement for oral anticoagulants before Day 30.
9. CRUSADE bleeding risk score >40.
10. Suspected aortic dissection.
11. History of gastrointestinal or genitourinary bleeding within the previous 3 months.
12. Refusal to receive blood transfusion if needed during the study.
13. Major surgery in the last month.
14. History of heparin-induced thrombocytopenia and bleeding diathesis.
15. Severe uncontrolled hypertension.
16. Prior (within 30 days prior to enrollment) or planned administration of thrombolytics, glycoprotein IIb/IIIa inhibitors, bivalirudin, or fondaparinux for the index MI.
17. Known relevant hematological deviations: hemoglobin (male) < 11 g/dL, hemoglobin (female) < 10 g/dL, hematocrit < 35%, platelet count < 100,000 cells/µL.
18. Use of Coumadin derivatives and/or Factor Xa inhibitor drugs within the last 7 days.
19. Chronic therapy with non-steroidal anti-inflammatory drugs (NSAIDs; except aspirin) , cyclooxygenase (COX)-2 inhibitors within 1 month before screening.
20. Known malignancies or other comorbid conditions with life expectancy < 1 year.
21. Known severe liver disease (i.e., aspartate aminotransferase [AST], alanine aminotransferase [ALT] > 3 × ULN).
22. Known positive serology for hepatitis B & C, HIV screen.
23. Known chronic kidney disease with estimated glomerular filtration rate (eGFR) <30 mL/min and/or dialysis.
24. Known allergy or intolerance to aspirin, clopidogrel, ticagrelor, prasugrel, bivalirudin, unfractionated heparin, P2Y12 antagonists, or contrast.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
To determine the safe and well tolerated dose of MT1002 in patients with ACS with NSTEMI and PCI. | 30 days
  Co-Primary endpoints:
  The number of patients with target ACT (200 -300 seconds [sec]) achieved on MT1002 (no switch to standard of care) prior/during PCI and PCI success.
  Adverse event (AE) of interest: bleeding events major (Bleeding Academic Research Consortium [BARC] Type 3-5)

SECONDARY OUTCOMES:
Major adverse cardiovascular event(s) | 30 days
To evaluate the anti-coagulation effect of MT1002 by activated partial thromboplastin time (aPTT) and activated clotting time (ACT) | 30 days
  Coagulation parameters (ACT, aPTT, PT, TT, FIB, INR) and Percentage of patients who achieve ACT ≥ 200 sec
To evaluate the anti-platelet effect of MT1002 by platelet aggregation (PA) | 30 days
  PA

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health - BMH, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: No